CLINICAL TRIAL: NCT03858010
Title: Validation of a Patient-reported Outcome Measurement Tool
Brief Title: Personalised Outcomes in Children With Recurrent Wheeze
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Imperial College Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 226984
Record Dates: First submitted 2019-02-26; First posted 2019-02-28 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Asthma in Children
Keywords: asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Wheeze and me questionnaire — validation of questionnaire assessing disease control and quality of life in preschool children with recurrent wheeze

SUMMARY:
This project aims to develop a PROM for preschool children with recurrent wheeze. Nearly one third of children will have at least one episode of wheeze in the first five years of life. The majority of these children grow out of the condition in early school years. However, their families go through challenging times often with numerous emergency department admissions and hospitalizations. Hospital admission rates for preschool children with wheeze attacks remain high and are increasing in the UK. New treatments have become available, but although current treatments speed recovery from a wheeze attack, still many children visit hospitals for rescue medications and medical reviews. Recent Australian data show that one fourth of these children remain at emergency departments for a less than four hours period, suggesting that with better information and education, these children could have remained at home.

Justification-Significance of the work By understanding what really matters for these families, clinicians and stakeholders will be better able to design interventions that will reduce the hospital attendances and admissions by empowering parents to manage their children's condition. More specifically, this tool will assist GPs identify which of these children need to be reviewed by specialists, aid holistic management, ensure interventions are meaningful for families and assess the benefits of novel treatments.

Methodology The items of the questionnaire have been generated through discussions with families in a qualitative research study conducted by the research team. These items will be refined and the questionnaire will be tested with families in different healthcare settings. Researchers will assess how well this questionnaire is identifying the children who present with greater number of hospital admissions and will be benefited from suggested interventions. The data will be analysed and based on the results, amendments will be made to the questionnaire, which can will then be introduced in the routine management of these children.

DETAILED DESCRIPTION:
The validation of the tool will take place at St Mary's Hospital.

The questionnaire aims to measure

1. incidence of wheeze attacks and use of rescue medications
2. parental/caregiver perception of recurrent wheeze control
3. parental/caregiver perception of effect of recurrent wheeze on family/child quality of life

Participants will be given the questionnaire at the emergency departments or outpatients clinics following having consented to the study and will be asked to fill in the questionnaire and return it to their clinician.

ELIGIBILITY:
Inclusion Criteria:

In this study caregivers of preschool children presenting with the second or more episode of wheeze that requires physician review with or without treatment (as per BTS definition of wheeze attack in preschool years) will be included.

Exclusion Criteria:

This study will exclude caregivers who do not consent to complete the questionnaire and therefore participate in the study.

This study will exclude caregivers of preschool children who present with their first episode of wheeze.

This study will exclude caregivers of preschool children who present with respiratory distress of any other etiology (foreign body inhalation, croup, lower respiratory tract infection, bronchiectasis, exacerbation of cystic fibrosis or ciliopathy)

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A total number of 350 parents of preschool children with recurrent wheeze will complete a questionnaire that assesses disease control and quality of life
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-08-13 (Actual); Primary Completion 2022-06-01 (Estimated); Study Completion 2022-06-05 (Estimated)

PRIMARY OUTCOMES:
feasibility of preschool wheeze assessment tool | March 2019 - March 2020
  how easily the questionnaire can be completed
content validity of the questionnaire | March 2019-March 2020
  assessing validity of each item of the questionnaire as comparing with item of already existing questionnaire

SECONDARY OUTCOMES:
reduction of avoidable emergency department admissions | March 2020-March 2021
  effect of the tool on number of avoidable emergency department presentations

CONTACTS AND LOCATIONS:
Overall Officials: Mando Watson, Principal Investigator — Imperial College Healthcare NHS Trust
Locations (1):
- St Mary's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
individual participant data will be anonymised and when anonymised can then be used by other researchers in the team

REFERENCES:
- [Background] Makrinioti H, Klaber R, Watson M. Around the world: preschool wheeze. Lancet Respir Med. 2017 Sep;5(9):688-689. doi: 10.1016/S2213-2600(17)30314-4. No abstract available. PMID 28853398